CLINICAL TRIAL: NCT05616273
Title: Stimulated Glucagon as a Biomarker of Hypoglycemic Risk in Type 1 Diabetes
Acronym: MUGGLE
Status: Completed | Type: Observational
Sponsor: University of Exeter (Other)
Collaborators: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-22-59; 319581 (Other: Health Research Authority); 22/LO/0719 (Other: Research Ethics Committee); Grant # 2012-04188 (Other: The Leona M. and Harry B. Helmsley Charitable Trust)
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: type 1 diabetes; autoimmune diabetes; beta cell destruction; hypoglycaemia; hyperglycaemia; glucagon; type 1 diabetes genetic risk; alpha cell
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma, RNA, PBMCs at serial timepoints after a meal or intravenous stimulus.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MMTT Visit 1, AST Visit 2: Mixed Meal Tolerance Test (MMTT) Visit 1 and Arginine Stimulated Test (AST) Visit 2
  Interventions: Other: Mixed Meal Tolerance Test (MMTT); Other: Arginine Stimulation Test (AST); Other: Home Finger Prick Sample
- AST Visit 1, MMTT Visit 2: Arginine Stimulated Test (AST) Visit 1 and Mixed Meal Tolerance Test (MMTT) Visit 2
  Interventions: Other: Mixed Meal Tolerance Test (MMTT); Other: Arginine Stimulation Test (AST); Other: Home Finger Prick Sample

INTERVENTIONS:
Other: Mixed Meal Tolerance Test (MMTT) — At either Visit 1 or Visit 2, participants will be given Ensure HP or Fortisip (a drink containing the same amounts of carbohydrates, protein and fats as there would be in a meal; 6ml/kg to a max of 360mls), and have blood samples collected, to measure insulin (C-peptide), glucose, and glucagon, at specific intervals: -10, 0, 30, 60, 90, 120 minutes post meal. This test is used to measure how a participant's beta cells are working to produce insulin after a meal and to check for reactive hypoglycaemia.
Other: Arginine Stimulation Test (AST) — At either Visit 1 or Visit 2, and Visit 3, participants will be given a dose of Arginine Hydrochloride (5 g Arginine during 1 min) by intravenous injection, and have blood samples collected to measure insulin (C-peptide), glucose, and glucagon, at specific intervals: -10, 0, 2, 5, 10, 15 and 30 minutes following the Arginine bolus injection. This test is designed primarily to test the maximum insulin secretion capacity of a participant's beta cells.
Other: Home Finger Prick Sample — Participants will be provided with a kit to collect an optional home finger prick sample the day after each visit, and return the sample using the prepaid addressed padded envelope provided.

SUMMARY:
Type 1 diabetes (T1D) results from destruction of insulin producing beta cells by the body's own immune system (autoimmunity) causing an individual to lose the ability to make enough insulin to control their blood sugar levels and need to have insulin injections to lower blood glucose levels. Whilst high blood sugar level is a problem for people with Type 1 diabetes, taking insulin medication to lower sugar levels, delayed meals and exercise can all result in dangerously low blood sugar levels (hypoglycaemia). The biological causes of hypoglycaemia, and ways to prevent it are poorly understood. In non-diabetic individuals, a hormone called glucagon is secreted naturally to raise blood glucose levels but it is unclear why glucagon secretion is impaired during hypoglycaemia in individuals with T1D.

The aim of this prospective observational study is to test the relationship between a glucagon stimulation test and risk of hypoglycaemia in T1D. It is hoped this research will establish whether this relationship could be used as a blood test and be a clinically useful biomarker of hypoglycaemia risk and, therefore, directly inform clinical care of people with T1D, particularly those with highest risk of hypoglycaemia.

Assessment of beta cell decline has traditionally relied on timed C-peptide measures following a standardised liquid meal known as the mixed meal tolerance test (MMTT). Home finger prick blood spot C-peptide measurement might be a practical, cheap, and non-invasive alternative to a MMTT and would allow regular assessment of beta cell function over time. If proven that this sample type is a robust alternative to the gold standard MMTT venous C-peptide, it would dramatically decrease the cost and participant burden of T1D research into beta cell function.

DETAILED DESCRIPTION:
Blood glucose levels are normally controlled by insulin, a hormone that lowers high blood glucose levels, and glucagon which is released into the blood to raise glucose when levels are low. For people with Type 1 diabetes (T1D), taking insulin medication to lower glucose levels can sometimes result in dangerously low blood sugar levels (hypoglycaemia). The ability to release glucagon and correct blood glucose can vary, particularly in people who have had T1D for years. The study aims to find out how blood glucagon levels after a stimulus compare to a person's own experience of hypoglycaemia, and hypoglycaemia. This research will establish whether glucagon measured after a meal could be used as a blood marker of hypoglycaemia risk and help to identify individuals at high risk.

Hypothesis: Low post-mixed meal (MM) stimulated glucagon secretion predicts hypoglycaemia.

Prior to consent, all potential participants will be provided with detailed written information about the study (that complies with the UK General Data Protection Regulation (GDPR) and Data Protection Act 2018) and an opportunity to discuss it with one of the research team. All participants will be informed of their right to withdraw from the study at any time without prejudice or jeopardy to any future clinical care.

A unique study ID will be allocated to the participant to link all participant study information and samples. The participant's clinical characteristics and sample results will be recorded on the participant's Case Report Form and entered on the study database.

All participants will undergo core data collection, measurements and provide fasted and stimulated blood samples via a cannula at the baseline MMTT and AST visits 1 and 2 and again at the 6 months 'Light MMTT' / repeat AST visit. The order of MMTT and AST tests in visits 1 and 2 will be randomised to check for an order effect. Test choice for Visit 3 depends on the peak glucagon results from Visits 1 and 2. At Visits 1 and 3, participants will be asked to complete the hypoglycaemia questionnaire data (Clarke and Gold scores) to assess awareness of hypoglycaemia and quality of life measures which may relate to the MM-glucagon. Participants will be given an Abbot FreeStyle Libre Pro continuous blood glucose monitor (CGM) and asked to perform a 2-week continuous measure of blood glucose (CGM). Clinical diabetes care will not be changed and participants with T1D will use their own insulin regimes and self-monitoring (even if CGM or Abbot FreeStyle Libre Pro) during the study.

Fasted samples will be obtained for baseline measures: routine glucose and HbA1c, plasma and serum for storage and future batched analysis including measures of glucose, glucagon, insulin (C-peptide) and other markers of interest, plus sodium heparin and PAXgenesRNA samples for T1D immune function analysis.

Stimulated samples (see test descriptions below): insulin (C-peptide), glucose and glucagon will be measured at all time points.

At the end of each test period, the participant's blood glucose will be checked and appropriate advice will be given relating to insulin dosage adjustments and a light meal will be provided.

A) Mixed Meal Tolerance Test (MMTT) at Visit 1 or 2 (approx 2½ hours) Rationale: The MMTT will provide confirmatory analysis of post-mixed meal glucagon stored in BD P800 and EDTA plasma samples at a range of standard MMTT time points (0, 30, 60, 90 and 120 min) in 75 people. Glucose will be measured in Fluoride Oxalate samples at the same time points.

Participants will:

* be monitored closely throughout their visit for any discomfort or problems and appropriate advice/support will be given if required.
* be given Ensure HP or Fortisip (6ml/kg to a max of 360mls)
* have blood samples collected, to measure insulin, C-peptide, glucose, and glucagon, at specific intervals: -10, 0, 30, 60, 90, 120 minutes post meal.

B) Arginine Stimulation Test (AST) Visit 1 or 2, and Visit 3 (approx 1 hour) Rationale. An MMTT (despite being convenient because it avoids the need for an IV stimulus) has limitations, including differences in gastric emptying, uptake and effects on enteroendocrine secretion. Therefore, responses will be compared during the MMTT with those obtained during an intravenous arginine challenge, Arginine Stimulation Test (AST), (5 g Arginine during 1 min) at a separate visit from the MMTT visit. Glucose, plasma glucagon and C-peptide will be measured at baseline and specific intervals following the Arginine bolus injection. This test is designed primarily to test the maximum insulin secretion capacity of a participant's beta cells.

The AST test involves:

* Set up. Intravenous catheters will be inserted into antecubital veins in both arms. One arm will be used for infusion of Arginine (amino acid), and the other arm for intermittent sampling.
* Baseline samples will be taken at -10 and 0 minutes. A maximally stimulating dose of Arginine Hydrochloride (5 g) will be injected intravenously for 45s. Samples will be collected at 2, 5, 10, 15 and 30 minute intervals following the Arginine bolus.

C) Home Finger Prick Sample (optional) - collected at home the day after each visit and returned to the research team, using pre-paid packaging provided.

Data Collection and Recording: Data will be initially recorded using a study-specific case report form (CRF), with hard copies stored in the Trial Master File (TMF). Anonymised research data will be recorded on a study-specific database and reviewed for discrepancies and missing data prior to analysis.

End of Study Definition: The end of the study is 8 months after the final participant's Visit 3 to allow for final collection of data.

Criteria for premature withdrawal from the study: Where a participant withdraws, data will be collected up to the point of withdrawal in line with the protocol and study SOPs. Where a participant has prematurely withdrawn but not revoked consent, data and samples will remain within the study and included in any analysis. Where consent is withdrawn, study samples and data will be kept/destroyed as per local guidelines.

Samples: A detailed SOP/work instruction will detail the clinical procedure for sample collection, labelling, logging and management. Central laboratory analysis of the study samples will be undertaken at the Exeter Blood Sciences Laboratory.

Stored samples: Surplus samples for storage should be processed, logged and frozen at -80°C within 24 hours of receipt. All saved samples will be stored under the study ID, with the file linking the study code to personal identifiable information held securely by the Principal Investigator, accessible only to personnel with training in data protection who require this information to perform their duties.

Safety, Definitions and Reporting:

Risks: The blood samples will be collected by members of the research team trained in venepuncture. During the MMTT/AST test, there is a possible risk of hyperglycaemia and appropriate advice/support will be given if required.

Benefits: The study may improve understanding of participants' hypoglycaemia risk. In the longer term, this work may provide evidence that the ability of alpha cells to release glucagon after a mixed meal is variable within people with T1D, associated with hypoglycaemia risk, and could be a biomarker for hypoglycaemia risk. Testing a blood spot assay for C-peptide on home finger prick samples may enable regular assessment of beta cell function without the need for patients/research participants to visit a healthcare/research centre which could revolutionise future diabetes care and research.

Definitions and reporting of adverse effects:

The timeframe for recording SAEs will be from the time of consent to one week following the last visit of a study subject. Any reportable adverse effects noted will be reported within 24 hours to the CI and the Sponsor as per standard NHS R&D protocols.

Insurance: Sponsor's public liability will be provided by the University of Exeter for the design and management of the study. NHS indemnity will apply for the conduct of the study at the site.

Data Handling & Record Keeping: The CI is responsible for ensuring that participant anonymity is protected and maintained, ensuring that their identities are protected from any unauthorised parties. The CI is the 'Custodian' of the data. All information related to study participants will be kept confidential and managed in accordance with the UK GDPR and Data Protection Act 2018, NHS Caldicott Guardian, UK Policy Framework for Health & Social Care, and Research Ethics Committee Approval.

A unique Study ID will be allocated to each participant. All study data and samples will be pseudo-anonymised and stored under the Study ID on a secure password-protected study database. Identifiable information will be stored on a separate, secure password-protected database held on an NHS server to enable the research team to undertake the study.

All paper copies of study data will be stored under ID number and kept in locked, access-controlled offices within the research facilities; research data will be held separately to identifiable information. Researchers involved in data analysis will not have access to personal identifiable data, only the anonymised research data. No identifiable data will be included in research publications or progress reports.

Any participant information required to be sent to a third party will adhere to these pseudo-anonymised parameters. No participant identifiable data will be sent outside the EU.

Record Retention and Archiving: When the research study is complete, it is a requirement of the UK Policy Framework for Health & Social Care and Sponsor Trust Policy that the records are kept for a further 15 years. At the end of the study, anonymised data will be included in the study's final dataset and stored indefinitely on vivli.org or similar sponsor/funder approved data repository. Personal data will be stored where consent is given by the participant to be contacted for follow-up on their future health status, and/or about participating in future studies. Where consent is given by the participant, their samples and data from the project will be gifted to the Peninsula Research Bank (an approved tissue bank, REC ref 19/SW/1059) to be used for future research.

At the end of the study, it will be archived by the CI at the University of Exeter.

Statistical analysis: For a sample size of 75, it should be possible to detect a correlation between stimulated glucagon and hypoglycaemia of r=0.3, with 95% confidence intervals 0.08 to 0.49, plus correlation of MM-induced increases in plasma glucagon to plasma co-peptin.

Compliance: The CI will ensure that the study is conducted in compliance with the principles of the Declaration of Helsinki (2013), the principles of GCP and in accordance with all applicable regulatory requirements including but not limited to the UK Policy Framework for Health & Social Care and the Medicines for Human Use (Clinical Trial) Regulations 2004, as amended in 2006, 2008 and 2009 and any future relevant or replacement EU Regulations, Trust and R&D Office policies and procedures and any subsequent amendments.

Publication Policy: Results will be written up and submitted for publication in a peer-reviewed journal(s). Abstracts will be submitted to national and international conferences. Results will be presented to clinical colleagues at regular in-house meetings. A letter/newsletter outlining the key findings of the study will be sent to all participants and will be uploaded to the study website. An in-person/online event may also be arranged.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 1 diabetes
* Insulin treated
* Known urine C-peptide status (using Urinary C-Peptide Creatinine Ratio [UCPCR], positive/negative defined by UCPCR 0.2nmol/mmol cut-off)
* Age 16-65 years inclusive
* Able and willing to provide informed consent/assent.

Exclusion Criteria:

* Age less than 16 year or over 65 years
* Pregnant or lactating (as this may limit blood sampling and affect T cell function)
* Any medical condition that, in the opinion of the investigator, would affect the safety of the subject's participation, or validity of results.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 75 individuals with long duration T1D, identified from participation in the TIGI study (UK IRAS ID: 141756, REC Number: 13/SW/0312), with consent to be contacted for future research.
  The TIGI participants have a clinical diagnosis of T1D, were on insulin from diagnosis and, if BMI was >30, were autoantibody positive. We will aim to recruit 50 people with undetectable C-peptide and 25 with detectable C-peptide. The selection of people with absent C-peptide allows a secondary analysis focussed on stimulated glucagon without any potential interaction with endogenous insulin secretion. It also focusses on a group of people known to be at high hypoglycaemia risk due to lack of endogenous insulin.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
A description of the strength and reproducibility of the relationship of post-Mixed Meal and Arginine stimulated glucagon with hypoglycaemia. | 22 months
  The longitudinal stability of stimulated glucagon will be described, including its relationship with variation in hypoglycaemia frequency, and the potential to predict future hypoglycaemia. This will be be determined from post-MM & Arginine-induced plasma glucagon levels, continuous glucose monitoring (CGM) time spent in hypoglycaemia, and self-reported hypoglycaemia episodes, hypoglycaemia fear/awareness, and fear of hypoglycaemia.

SECONDARY OUTCOMES:
Longitudinal variability of glucagon levels and its relationship to episodes of hypoglycaemia in long-duration T1D. | 22 months
  Stimulated and plasma glucagon levels, and continuous glucose monitoring (CGM) will be used to describe longitudinal variability of glucagon levels and its relationship to episodes of hypoglycaemia in long-duration T1D.
The relationship between plasma glucagon levels under basal conditions, following a stimulation (by mixed meal or arginine) | 22 months
  A mechanistic understanding of the relationship between plasma glucagon levels under basal conditions, following a stimulation (by mixed meal or arginine) will be derived. The cause/effect relationship between hypoglycaemia and alpha cell function will be investigated via stimulated and plasma glucagon levels, and continuous glucose monitoring (CGM).
Home finger prick blood spot C-peptide measurement is a practical alternative to MMTT | 22 months
  Establish if home finger prick blood spot C-peptide measurement is a practical alternative to MMTT by comparison of C-peptide levels in capillary blood spot samples to levels in samples collected during a 'gold standard' MMTT.

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Oram, MRCP (neph), Principal Investigator — University of Exeter
Locations (1):
- Royal Devon University Healthcare NHS Foundation Trust, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The study's final anonymised dataset will be uploaded to vivli.org, a sponsor/funder approved data repository by October 2026. In addition, where consent is given by the participant, their samples and data from the project will be gifted to the Peninsula Research Bank (an approved tissue bank, REC ref 19/SW/1059) in Exeter to be used for future research.
  Any participant information required to be sent to a third party will adhere to these pseudo-anonymised parameters, this includes the participant's date of birth, gender, and unique study ID. No participant identifiable data will be sent outside the EU.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available 12 months after the study end.
Access Criteria: Applications submitted via the approved data repository would be considered.

REFERENCES:
- [Background] Lund A, Bagger JI, Wewer Albrechtsen NJ, Christensen M, Grondahl M, Hartmann B, Mathiesen ER, Hansen CP, Storkholm JH, van Hall G, Rehfeld JF, Hornburg D, Meissner F, Mann M, Larsen S, Holst JJ, Vilsboll T, Knop FK. Evidence of Extrapancreatic Glucagon Secretion in Man. Diabetes. 2016 Mar;65(3):585-97. doi: 10.2337/db15-1541. Epub 2015 Dec 15. PMID 26672094
- [Result] Gerich JE, Langlois M, Noacco C, Karam JH, Forsham PH. Lack of glucagon response to hypoglycemia in diabetes: evidence for an intrinsic pancreatic alpha cell defect. Science. 1973 Oct 12;182(4108):171-3. doi: 10.1126/science.182.4108.171. PMID 4581053
- [Result] Frier BM. Hypoglycaemia in diabetes mellitus: epidemiology and clinical implications. Nat Rev Endocrinol. 2014 Dec;10(12):711-22. doi: 10.1038/nrendo.2014.170. Epub 2014 Oct 7. PMID 25287289
- [Result] Hypoglycemia in the Diabetes Control and Complications Trial. The Diabetes Control and Complications Trial Research Group. Diabetes. 1997 Feb;46(2):271-86. PMID 9000705
- [Result] Epidemiology of severe hypoglycemia in the diabetes control and complications trial. The DCCT Research Group. Am J Med. 1991 Apr;90(4):450-9. PMID 2012085
- [Result] Cryer PE. Minireview: Glucagon in the pathogenesis of hypoglycemia and hyperglycemia in diabetes. Endocrinology. 2012 Mar;153(3):1039-48. doi: 10.1210/en.2011-1499. Epub 2011 Dec 13. PMID 22166985
- [Result] Rorsman P, Ramracheya R, Rorsman NJ, Zhang Q. ATP-regulated potassium channels and voltage-gated calcium channels in pancreatic alpha and beta cells: similar functions but reciprocal effects on secretion. Diabetologia. 2014 Sep;57(9):1749-61. doi: 10.1007/s00125-014-3279-8. Epub 2014 Jun 7. PMID 24906950
- [Result] Bollyky J, Greenbaum CJ. Editorial: The role of glucagon in postprandial hyperglycemia--the jury's still out. J Clin Endocrinol Metab. 2007 Aug;92(8):2879-81. doi: 10.1210/jc.2007-1312. No abstract available. PMID 17682088
- [Result] Zenz S, Mader JK, Regittnig W, Brunner M, Korsatko S, Boulgaropoulos B, Magnes C, Raml R, Narath SH, Eller P, Augustin T, Pieber TR. Impact of C-Peptide Status on the Response of Glucagon and Endogenous Glucose Production to Induced Hypoglycemia in T1DM. J Clin Endocrinol Metab. 2018 Apr 1;103(4):1408-1417. doi: 10.1210/jc.2017-01836. PMID 29408994
- [Result] Brissova M, Haliyur R, Saunders D, Shrestha S, Dai C, Blodgett DM, Bottino R, Campbell-Thompson M, Aramandla R, Poffenberger G, Lindner J, Pan FC, von Herrath MG, Greiner DL, Shultz LD, Sanyoura M, Philipson LH, Atkinson M, Harlan DM, Levy SE, Prasad N, Stein R, Powers AC. alpha Cell Function and Gene Expression Are Compromised in Type 1 Diabetes. Cell Rep. 2018 Mar 6;22(10):2667-2676. doi: 10.1016/j.celrep.2018.02.032. PMID 29514095
- [Result] Brown RJ, Sinaii N, Rother KI. Too much glucagon, too little insulin: time course of pancreatic islet dysfunction in new-onset type 1 diabetes. Diabetes Care. 2008 Jul;31(7):1403-4. doi: 10.2337/dc08-0575. PMID 18594062
- [Result] Sherr J, Tsalikian E, Fox L, Buckingham B, Weinzimer S, Tamborlane WV, White NH, Arbelaez AM, Kollman C, Ruedy KJ, Cheng P, Beck RW; Diabetes Research in Children Network. Evolution of abnormal plasma glucagon responses to mixed-meal feedings in youth with type 1 diabetes during the first 2 years after diagnosis. Diabetes Care. 2014 Jun;37(6):1741-4. doi: 10.2337/dc13-2612. Epub 2014 Apr 2. PMID 24696460
- [Result] Orskov C, Wettergren A, Holst JJ. Secretion of the incretin hormones glucagon-like peptide-1 and gastric inhibitory polypeptide correlates with insulin secretion in normal man throughout the day. Scand J Gastroenterol. 1996 Jul;31(7):665-70. doi: 10.3109/00365529609009147. PMID 8819215
- [Result] Rickels MR, Evans-Molina C, Bahnson HT, Ylescupidez A, Nadeau KJ, Hao W, Clements MA, Sherr JL, Pratley RE, Hannon TS, Shah VN, Miller KM, Greenbaum CJ; T1D Exchange beta-Cell Function Study Group. High residual C-peptide likely contributes to glycemic control in type 1 diabetes. J Clin Invest. 2020 Apr 1;130(4):1850-1862. doi: 10.1172/JCI134057. PMID 31895699
- [Result] Zhang Q, Ramracheya R, Lahmann C, Tarasov A, Bengtsson M, Braha O, Braun M, Brereton M, Collins S, Galvanovskis J, Gonzalez A, Groschner LN, Rorsman NJ, Salehi A, Travers ME, Walker JN, Gloyn AL, Gribble F, Johnson PR, Reimann F, Ashcroft FM, Rorsman P. Role of KATP channels in glucose-regulated glucagon secretion and impaired counterregulation in type 2 diabetes. Cell Metab. 2013 Dec 3;18(6):871-82. doi: 10.1016/j.cmet.2013.10.014. PMID 24315372
- [Result] Porksen S, Nielsen LB, Kaas A, Kocova M, Chiarelli F, Orskov C, Holst JJ, Ploug KB, Hougaard P, Hansen L, Mortensen HB; Hvidore Study Group on Childhood Diabetes. Meal-stimulated glucagon release is associated with postprandial blood glucose level and does not interfere with glycemic control in children and adolescents with new-onset type 1 diabetes. J Clin Endocrinol Metab. 2007 Aug;92(8):2910-6. doi: 10.1210/jc.2007-0244. Epub 2007 May 22. PMID 17519307
- [Result] Hare KJ, Vilsboll T, Holst JJ, Knop FK. Inappropriate glucagon response after oral compared with isoglycemic intravenous glucose administration in patients with type 1 diabetes. Am J Physiol Endocrinol Metab. 2010 Apr;298(4):E832-7. doi: 10.1152/ajpendo.00700.2009. Epub 2010 Jan 26. PMID 20103744
- [Result] Marren SM, Hammersley S, McDonald TJ, Shields BM, Knight BA, Hill A, Bolt R, Tree TI, Roep BO, Hattersley AT, Jones AG, Oram RA; TIGI consortium. Persistent C-peptide is associated with reduced hypoglycaemia but not HbA1c in adults with longstanding Type 1 diabetes: evidence for lack of intensive treatment in UK clinical practice? Diabet Med. 2019 Sep;36(9):1092-1099. doi: 10.1111/dme.13960. Epub 2019 Jun 27. PMID 30955221
- [Result] Geddes J, Wright RJ, Zammitt NN, Deary IJ, Frier BM. An evaluation of methods of assessing impaired awareness of hypoglycemia in type 1 diabetes. Diabetes Care. 2007 Jul;30(7):1868-70. doi: 10.2337/dc06-2556. Epub 2007 Apr 6. No abstract available. PMID 17416785
- [Result] Wewer Albrechtsen NJ, Bak MJ, Hartmann B, Christensen LW, Kuhre RE, Deacon CF, Holst JJ. Stability of glucagon-like peptide 1 and glucagon in human plasma. Endocr Connect. 2015 Mar;4(1):50-7. doi: 10.1530/EC-14-0126. Epub 2015 Jan 16. PMID 25596009
- [Result] Atkinson MA, Leiter EH. The NOD mouse model of type 1 diabetes: as good as it gets? Nat Med. 1999 Jun;5(6):601-4. doi: 10.1038/9442. No abstract available. PMID 10371488
- [Result] Chen YG, Mathews CE, Driver JP. The Role of NOD Mice in Type 1 Diabetes Research: Lessons from the Past and Recommendations for the Future. Front Endocrinol (Lausanne). 2018 Feb 23;9:51. doi: 10.3389/fendo.2018.00051. eCollection 2018. PMID 29527189
- [Result] Ramracheya R, Ward C, Shigeto M, Walker JN, Amisten S, Zhang Q, Johnson PR, Rorsman P, Braun M. Membrane potential-dependent inactivation of voltage-gated ion channels in alpha-cells inhibits glucagon secretion from human islets. Diabetes. 2010 Sep;59(9):2198-208. doi: 10.2337/db09-1505. Epub 2010 Jun 14. PMID 20547976
- [Result] Rorsman P, Ashcroft FM. Pancreatic beta-Cell Electrical Activity and Insulin Secretion: Of Mice and Men. Physiol Rev. 2018 Jan 1;98(1):117-214. doi: 10.1152/physrev.00008.2017. PMID 29212789
- [Result] McDonald TJ, Perry MH, Peake RW, Pullan NJ, O'Connor J, Shields BM, Knight BA, Hattersley AT. EDTA improves stability of whole blood C-peptide and insulin to over 24 hours at room temperature. PLoS One. 2012;7(7):e42084. doi: 10.1371/journal.pone.0042084. Epub 2012 Jul 30. PMID 22860060
- [Result] McDonald TJ, Besser RE, Perry M, Babiker T, Knight BA, Shepherd MH, Ellard S, Flanagan SE, Hattersley AT. Screening for neonatal diabetes at day 5 of life using dried blood spot glucose measurement. Diabetologia. 2017 Nov;60(11):2168-2173. doi: 10.1007/s00125-017-4383-3. Epub 2017 Aug 5. PMID 28779213
- [Result] Battelino T, Danne T, Bergenstal RM, Amiel SA, Beck R, Biester T, Bosi E, Buckingham BA, Cefalu WT, Close KL, Cobelli C, Dassau E, DeVries JH, Donaghue KC, Dovc K, Doyle FJ 3rd, Garg S, Grunberger G, Heller S, Heinemann L, Hirsch IB, Hovorka R, Jia W, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Levine B, Mayorov A, Mathieu C, Murphy HR, Nimri R, Norgaard K, Parkin CG, Renard E, Rodbard D, Saboo B, Schatz D, Stoner K, Urakami T, Weinzimer SA, Phillip M. Clinical Targets for Continuous Glucose Monitoring Data Interpretation: Recommendations From the International Consensus on Time in Range. Diabetes Care. 2019 Aug;42(8):1593-1603. doi: 10.2337/dci19-0028. Epub 2019 Jun 8. PMID 31177185
- [Result] Milan AM, D'Souza RF, Pundir S, Pileggi CA, Thorstensen EB, Barnett MP, Markworth JF, Cameron-Smith D, Mitchell CJ. Older Adults Have Delayed Amino Acid Absorption after a High Protein Mixed Breakfast Meal. J Nutr Health Aging. 2015 Oct;19(8):839-45. doi: 10.1007/s12603-015-0500-5. PMID 26412288
- [Result] Salehi A, Gunnerud U, Muhammed SJ, Ostman E, Holst JJ, Bjorck I, Rorsman P. The insulinogenic effect of whey protein is partially mediated by a direct effect of amino acids and GIP on beta-cells. Nutr Metab (Lond). 2012 May 30;9(1):48. doi: 10.1186/1743-7075-9-48. PMID 22647249
- [Result] De Marinis YZ, Salehi A, Ward CE, Zhang Q, Abdulkader F, Bengtsson M, Braha O, Braun M, Ramracheya R, Amisten S, Habib AM, Moritoh Y, Zhang E, Reimann F, Rosengren A, Shibasaki T, Gribble F, Renstrom E, Seino S, Eliasson L, Rorsman P. GLP-1 inhibits and adrenaline stimulates glucagon release by differential modulation of N- and L-type Ca2+ channel-dependent exocytosis. Cell Metab. 2010 Jun 9;11(6):543-553. doi: 10.1016/j.cmet.2010.04.007. PMID 20519125
- [Result] Winzeler B, Cesana-Nigro N, Refardt J, Vogt DR, Imber C, Morin B, Popovic M, Steinmetz M, Sailer CO, Szinnai G, Chifu I, Fassnacht M, Christ-Crain M. Arginine-stimulated copeptin measurements in the differential diagnosis of diabetes insipidus: a prospective diagnostic study. Lancet. 2019 Aug 17;394(10198):587-595. doi: 10.1016/S0140-6736(19)31255-3. Epub 2019 Jul 11. PMID 31303316
- [Result] Knudsen JG, Hamilton A, Ramracheya R, Tarasov AI, Brereton M, Haythorne E, Chibalina MV, Spegel P, Mulder H, Zhang Q, Ashcroft FM, Adam J, Rorsman P. Dysregulation of Glucagon Secretion by Hyperglycemia-Induced Sodium-Dependent Reduction of ATP Production. Cell Metab. 2019 Feb 5;29(2):430-442.e4. doi: 10.1016/j.cmet.2018.10.003. Epub 2018 Nov 8. PMID 30415925
- [Result] Walker JN, Ramracheya R, Zhang Q, Johnson PR, Braun M, Rorsman P. Regulation of glucagon secretion by glucose: paracrine, intrinsic or both? Diabetes Obes Metab. 2011 Oct;13 Suppl 1:95-105. doi: 10.1111/j.1463-1326.2011.01450.x. PMID 21824262
- [Result] Vergari E, Knudsen JG, Ramracheya R, Salehi A, Zhang Q, Adam J, Asterholm IW, Benrick A, Briant LJB, Chibalina MV, Gribble FM, Hamilton A, Hastoy B, Reimann F, Rorsman NJG, Spiliotis II, Tarasov A, Wu Y, Ashcroft FM, Rorsman P. Insulin inhibits glucagon release by SGLT2-induced stimulation of somatostatin secretion. Nat Commun. 2019 Jan 11;10(1):139. doi: 10.1038/s41467-018-08193-8. PMID 30635569
- [Result] Ramracheya RD, McCulloch LJ, Clark A, Wiggins D, Johannessen H, Olsen MK, Cai X, Zhao CM, Chen D, Rorsman P. PYY-Dependent Restoration of Impaired Insulin and Glucagon Secretion in Type 2 Diabetes following Roux-En-Y Gastric Bypass Surgery. Cell Rep. 2016 May 3;15(5):944-950. doi: 10.1016/j.celrep.2016.03.091. Epub 2016 Apr 21. PMID 27117413
- [Result] Hamilton A, Zhang Q, Salehi A, Willems M, Knudsen JG, Ringgaard AK, Chapman CE, Gonzalez-Alvarez A, Surdo NC, Zaccolo M, Basco D, Johnson PRV, Ramracheya R, Rutter GA, Galione A, Rorsman P, Tarasov AI. Adrenaline Stimulates Glucagon Secretion by Tpc2-Dependent Ca2+ Mobilization From Acidic Stores in Pancreatic alpha-Cells. Diabetes. 2018 Jun;67(6):1128-1139. doi: 10.2337/db17-1102. Epub 2018 Mar 21. PMID 29563152